CLINICAL TRIAL: NCT01741402
Title: Effects of Training in a Virtual Environment on the Performance of Gait, Postural Control and Executive Functions in Healthy Elderly
Brief Title: Effects of Training in a Virtual Environment in Healthy Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Coordination for the Improvement of Higher Education Personnel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USPNEC004
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2012-11

CONDITIONS: Elderly
Keywords: Control posture; Gait; Virtual Reality; Elderly
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Virtual Reality Training (Experimental): The virtual reality training was done by experimental group with ten games of Nintendo Wii Fit.
  Interventions: Device: Virtual Reality Training
- Physical Therapy (Active Comparator): The Control Group was trained by conventional Physical Therapy exercises.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Device: Virtual Reality Training — The participants of the study trained 10 balance games during 14 sessions
  Arms: Virtual Reality Training
Other: Physical Therapy — Patients of the control group was trained with balance exercises.
  Arms: Physical Therapy

SUMMARY:
The objective of this work was to compare the effects of two balance training programs, one Nintendo Wii Fit-based and the other traditionally-based without the use of a gaming system, on the (1) balance, (2) gait, (3) functionality and (4) cognition ability in older adults. It is a prospective, single blinded, randomized clinical trial performed at Center of Research of the courses of Speech Therapy, Physical Therapy and Occupational Therapy of São Paulo University. Thirty-two older adults are randomly in control and experimental group, 16 each one. The study includes only participants scoring at least 24 in the Mini-Mental State Examination to rule out effects of dementia; without the presence of depression, according to the Geriatric Depression Scale of Yesaváge - version 15 (GDS-15 ≤ 5) and scores on the Berg Balance Scale (EBB ≥ 41).

DETAILED DESCRIPTION:
The objective of this work is to compare the effects of two balance training programs, one Nintendo Wii Fit-based and the other traditionally-based without the use of a gaming system, on balance, gait, functionality and cognition ability in older adults. It is a prospective, single blinded, randomized clinical trial performed at Center of Research of the courses of Speech Therapy, Physical Therapy and Occupational Therapy of São Paulo University. Thirty-two older adults are randomly in control and experimental group, 16 each one. Both groups performed 14 training sessions, twice a week, for seven weeks. Each session is composed of a 30 minute-global-exercise series including stretching, muscle strength and axial mobility exercises. After this, both groups performed more 30 minutes of balance training: the control group performed balance exercises without external cues, visual or auditory feedbacks or cognitive stimulations; the experimental group performed the balance training with 10 Wii Fit games which stimulated motor and cognitive functions. The main outcome measures are: (1) Mini-BESTest of Dynamic Balance Evaluation; (2) Dynamic Gait Index (DGI); (3) Montreal Cognitive Assessment (MoCA); and (4) Falls Efficacy Scale - International (FES-I).

ELIGIBILITY:
Inclusion Criteria:

* Age 60 to 85 years.
* Absence of other neurological disorders or co-morbidities that may affect gait;
* Absence of dementia (score above 24 on the Mini Mental State Examination - MMSE);
* Absence of depression (score above 5 on the Geriatric Depression Scale of Yesaváge - version 15);
* Score on the Berg Balance Scale above 41;
* Vision and hearing adequate or corrected to normal;
* Ability to walk independently;

Exclusion Criteria:

* Biomechanical alterations (other pathologies) that could compromise the completion of training;
* Presence of any neurological, auditory or visual deficit that could compromise distracting task performance during balance and gait training;

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-02; Primary Completion 2013-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Mini-BESTest of Dynamic Balance Evaluation - Balance Evaluation Systems Test | Up to 3 months
  The Mini-BESTest test is a 14-item test that focuses on dynamic balance, specifically anticipatory transitions, postural responses, sensory orientation and dynamic gait.

SECONDARY OUTCOMES:
Dynamic Gait Index | Up to 3 months
  The scale assesses the ability to adapt the gait during motor tasks with different demands.
Montreal Cognitive Assessment | Up to 3 months
  This scale was developed in order to detect mild degrees of cognitive impairment. The instrument assesses different cognitive domains such as attention and concentration, executive functions, memory, language, visuo-constructive skills, calculations, and orientation.
Falls Efficacy Scale - International | Up to 3 months
  The Falls Efficacy Scale-International (FES-I)measures the level of concern about falling during social and physical activities inside and outside the home whether or not the person actually does the activity.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elisa P Piemonte, PhD, Study Director — University of Sao Paulo; Keyte Guedes, MS Student, Principal Investigator — University of Sao Paulo; Alexandra M Lobo, MS Student, Principal Investigator — University of Sao Paulo
Locations (1):
- Center of Research of the courses of Speech Therapy, Physical Therapy and Occupational Therapy of São Paulo University, São Paulo, São Paulo, Brazil